CLINICAL TRIAL: NCT02338999
Title: The Role of PPAR-Gamma Agonists in Immunomodulation and Vascular Prevention in SLE (PPAR-SLE)
Brief Title: Role of PPAR-y Agonists in Immunomodulation and Vascular Prevention in SLE (PPAR-SLE)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 150060; 15-AR-0060
Record Dates: First submitted 2015-01-14; First posted 2015-01-15 (Estimated); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2020-07-14

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Autoimmunity Pathogenesis; Atherosclerosis; Adult
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Atherosclerosis | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pioglitazone, then placebo (Experimental): Treatment with pioglitazone up to 45 mg orally daily for three months. Followed by a two-month washout period before cross over to placebo orally daily for three months. A randomly selected subset of subjects underwent optional FDG-PET/CT for measurement of inflammatory activity in the blood vessels.
  Interventions: Radiation: PET/CT; Drug: Pioglitazone; Drug: Placebo
- Placebo, then Pioglitazone (Experimental): Treatment with placebo orally daily for three months. Followed by a two-month washout period before cross over to pioglitazone up to 45 mg daily orally for an additional three months. A randomly selected subset of subjects underwent optional FDG-PET/CT for measurement of inflammatory activity in the blood vessels.
  Interventions: Radiation: PET/CT; Drug: Pioglitazone; Drug: Placebo

INTERVENTIONS:
Radiation: PET/CT — The combined PET/CT scans provide images that pinpoint the anatomic location of abnormal metabolic activity within the body.
Drug: Pioglitazone — Increases insulin sensitivity in muscle and adipose tissue, and inhibits hepatic gluconeogenesis.
Drug: Placebo

SUMMARY:
Background:

- Lupus causes a person s immune system to attack the body. It can cause blood vessel problems, heart attack, or stroke. Researchers want to see if the drug pioglitazone may help.

Objectives:

- To see how well pioglitazone improves blood vessel function and decreases blood vessel inflammation. To study its effect on lupus symptoms.

Eligibility:

- Adults at least 18 years old with lupus.

Design:

* Participants will be screened with medical history, heart test, and blood and urine tests. They may have a bone density test.
* Visit 1:
* Participants will have:
* Physical exam and blood drawn.
* Peripheral Arterial Tonometry (Endopat). A cup will be placed on the finger and a pressure cuff on the arm.
* Cardio-ankle vascular index (CAVI) and/or Sphygmocor. Electrodes will be placed on both wrists, a microphone on the chest, and a blood pressure cuff on each arm and leg. Another test will involve placing a small device on a fingertip.
* 18-Fluorodeoxyglucose (FDG) positron emission tomography/computerized tomography (PET/CT) (some participants). A radioactive sugar will be injected into a small plastic tube in an arm vein. Participants will lie on a bed that moves in and out of a scanner that takes pictures.
* Participants will get a 3-month-supply of the study drug or placebo. After 1 week, their dose may increase.
* After those 3 months, they will not take either drug for 8 weeks. Then they will switch and take the other drug for 3 months.
* Participants will have 6 more visits over 8 months after Visit 1. Tests from Visit 1 may be repeated. They may have a urine test.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune disease of unclear cause that affects primarily women of childbearing age. Patients with lupus have a significantly increased risk of developing complications of their blood vessels due to accelerated hardening of the arteries (atherosclerosis). These complications include heart attacks and stroke. No drug to date has proven to prevent this type of complication in lupus and premature vascular disease significantly impacts the quality of life of these patients and enhances their risk of death.

The thiazolidinediones (TZD) are a class of drugs approved for the treatment of patients with type 2 diabetes mellitus (DM); they belong to the family of drugs that activate the peroxisome proliferator-activated receptor-gamma (PPAR-gamma). They have been proposed to have strong anti-atherogenic and anti-inflammatory effects even in patients without diabetes. Recent work from our group and others indicates that TZDs significantly improve vascular damage, dysfunction of blood vessels and disease activity in mouse models of lupus and abrogate atherosclerosis. We recently identified the TZD pioglitazone as an effective drug in modulation of vascular function and disease activity in patients with rheumatoid arthritis. In addition, we have found in mouse models of lupus and in in vitro experiments with human lupus cells, that pioglitazone has important roles in modulating immune function and vascular manifestations. Furthermore, this drug is not immunosuppressive, adding an additional advantage when compared to other medications used in this disease.

We propose that TZDs could significantly improve blood vessel function and play a role in atherosclerosis prevention in human SLE, in addition to modifying lupus disease activity. The major goal of the proposed research is to assess the effects of the PPAR-gamma agonist pioglitazone in SLE on vascular function and inflammation and on SLE disease activity. The results of the study may lead to the characterization of a new therapeutic target with dual effects on lupus and its associated blood vessel damage

ELIGIBILITY:
-INCLUSION CRITERIA:

1. For females and males 18 years old or older: females should be on adequate contraception if they are of child-bearing potential, which should be documented by a clinician, unless patients or their spouse/partner(s) have previously undergone a sterilization procedure. Adequate contraception will be considered:

   * Intrauterine device (IUD),
   * Hormone implants,
   * Injectable contraceptives,
   * Oral contraceptives plus a barrier method (male condom, female condom or diaphragm),
   * Abstinence, or
   * A vasectomized partner.
2. Meet revised ACR criteria and 2012 SLICC criteria for SLE and have: a) a baseline SLEDAI-2K greater than or equal to 4 and <20 or a clinical SLEDAI-2K greater than or equal to 2 (not considering anti-dsDNA or complement levels) and b) lack of BILAG A flare at baseline.
3. Stable doses of immunosuppressants and/or antimalarials for at least 3 months, and/or corticosteroids for at least 2 weeks. The prednisone dose may be increased after screening visit as long as the total dose is less than 20 mg of prednisone or equivalent per

   day and the subject is on stable dose for at least 2 weeks prior to their Day 1 visit. If on statins, should have been on stable doses for at least 6 months.
4. Allowed concomitant lupus-related medications

Antimalarials,

Prednisone greater than or equal to 20mg daily or equivalent doses of other corticosteroids;

Immunosuppressants:

* Mycophenolate mofetil, up to 3000 mg/day,
* Methotrexate, up to 30 mg/week,
* Azathioprine, up to 3 mg/kg/day,
* Leflunomide, up to 20 mg/day,
* Cyclosporine, up to 5 mg/kg/day
* Tacrolimus, up to 0.1 mg/kg/day

NSAIDS and aspirin

Note: While it would be highly desirable to maintain corticosteroid dosage at constant level for trial duration, it is impractical to anticipate that all patients with active SLE can be maintained without therapy modification for an 8-month period. Because corticosteroids are acceptable agents for treatment of the vast majority of minor lupus flares, and patients with major flares (BILAG 2004 A or recent change in medications) will be excluded, this will provide standardized treatment across study population that can be easily analyzed. An increase in prednisone dose of less than or equal to <10 mg/day from their prednisone dose at study entry will be permitted during the trial for increased disease activity with a standardized taper allowable in small monthly decrements to the patient s baseline dose or 5 mg/day, whichever is less.

EXCLUSION CRITERIA:

1. Pregnant or lactating women
2. Expected need for major surgery during trial.
3. Current or previous diagnosis of malignant disease, except for basal cell or squamous cell carcinoma of the skin with complete excision and clear borders or adequately treated in situ carcinoma of the cervix.
4. Acute infections identified during screening that require antibiotics. These subjects would be eligible to participate following resolution of infection before Day 1 visit within the allowed 46 days screening period. The subject will re-screen if it extends beyond the

   allowed 46 days screening period.
5. Chronic infections such as hepatitis B, hepatitis C, HIV or Tuberculosis.
6. Current use of cyclophosphamide or having received cyclophosphamide within the last year.
7. Prior history of hemorrhagic cystitis or hematuria while receiving cyclophosphamide that could not be explained by other causes.
8. Current use (within 3 months) of tocilizumab, rituximab, belimumab, intravenous gammaglobulin or other biologic.
9. History of poor compliance with medical care, study visits and/or medication use.
10. Receipt of any investigational new drug or device within 30 days prior to screening or 5 half-lives of the agent <TAB>(whichever is longer), or any investigational new drug with known long-term effects.
11. Pioglitazone is not recommended in patients with symptomatic heart failure. Patients with current heart failure (NYHA class II, III or IV) and/or a left ventricular ejection fraction of <45% by echocardiogram at screening will be excluded.
12. Significant impairment of major organ function (lung, heart, liver, kidney) or any condition that, in the opinion of the Investigator, would jeopardize the subject s safety following exposure to the study drug.
13. Known hypersensitivity to TZDs
14. Serum hepatic transaminase levels > 2 times upper normal limit, or clinical evidence of active liver disease at screening. The only exception is patients with confirmed non-alcoholic fatty liver disease (NAFLD) where pioglitazone has been reported to have a therapeutic role.
15. Diagnosis of DM or meeting DM criteria at screening visit, as established by new classification criteria: Patients with diabetes are excluded because diabetes by itself will induce profound changes in endothelial function and we want to assess the effects of PPAR agonists in vascular risk beyond changes in insulin resistance.
16. Known latex allergy for EndoPAT test
17. Patients with severe Raynaud's phenomenon, history of finger ulcers or finger gangrene will not undergo Endopat testing.
18. Patients with severe SLE at baseline, as quantified as SLEDAI-2K >20.
19. Patients with active lupus nephritis or active CNS lupus at baseline even if SLEDAI-2K <20. Active disease will be considered as CNS or renal disease that require aggressive immunosuppression. Active CNS disease will be diagnosed based on clinical presentation and physical exam, exclusion of other conditions that could explain symptomatology and, when warranted, ancillary tests (imaging) that support the diagnosis.

    Patients that are not on induction therapy for lupus nephritis and have chronic (more than 6 months), stable proteinuria <750 mg/gram in protein:creatinine ratio but otherwise considered to have no evidence of active lupus nephritis (e.g. no cellular casts and stable serum creatinine < 2 mg/dL) over the last 6 months, will be included in the study.

    In selected patients with potentially confounding clinical factors, consults will be requested to help clarify the nature of any underlying renal disease that may affect inclusion.
20. Postmenopausal women who have not undergone a DEXA scan over the last year will undergo a DEXA scan at screening. Patients with a better than -2.5 will be included. Postmenopausal women who have undergone a DEXA scan during the last year and have a T score better than -2.5 will be included without repeating the DEXA scan prior to enrollment. If the T score is worse than -2.5, they will be excluded from participating unless the subject is willing to begin appropriate treatment for osteoporosis by Visit Day 1. Postmenopausal women who have undergone a DEXA scan during the last year, have a T score worse than -2.5 and are not on bisphosphonates or other appropriate therapy will be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana J Kaplan, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Hasni S, Temesgen-Oyelakin Y, Davis M, Chu J, Poncio E, Naqi M, Gupta S, Wang X, Oliveira C, Claybaugh D, Dey A, Lu S, Carlucci P, Purmalek M, Manna ZG, Shi Y, Ochoa-Navas I, Chen J, Mukherjee A, Han KL, Cheung F, Koroleva G, Belkaid Y, Tsang JS, Apps R, Thomas DE, Heller T, Gadina M, Playford MP, Li X, Mehta NN, Kaplan MJ. Peroxisome proliferator activated receptor-gamma agonist pioglitazone improves vascular and metabolic dysfunction in systemic lupus erythematosus. Ann Rheum Dis. 2022 Oct 12;81(11):1576-1584. doi: 10.1136/ard-2022-222658. PMID 35914929
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-AR-0060.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 88 subjects were consented; 5 subjects declined participation after consent and 3 subjects did not meet eligibility criteria.
Groups:
- Pioglitazone, Then Placebo: Treatment with pioglitazone 45 mg daily (may be titrated down to 30 mg if subject experiences weight gain or other side effects) for three months. Followed by a two-month washout period before cross over to placebo treatment for 3 months.
- Placebo, Then Pioglitazone: Treatment with placebo for 3 months. Followed by a 2-month washout period before cross over to pioglitazone 45 mg daily (may be titrated down to 30 mg if subject experiences weight gain or other side effects) for an additional 3 months.
Period: First Intervention
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Started | 39 | 41
Completed | 36 | 40
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1
Period: Washout Period
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Started | 36 | 40
Completed | 36 | 38
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Second Intervention
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Started | 36 | 38
Completed | 36 | 36
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 39 | 72
  >=65 years | 6 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 37 | 70
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 17 | 33
  Not Hispanic or Latino | 22 | 24 | 46
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 17 | 17 | 34
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Vascular Function and Cardiometabolic Risk as Measured by Left CAVI at Month 3
Description: Change in vascular function using non-invasive vascular tests, measuring vascular compliance - Cardio ankle vascular index (CAVI).
  CAVI is an index reflecting the stiffness of the artery from the heart to ankles; it increases with atherosclerosis progression. CAVI was measured using VaSera-1500A (Fukuda Denshi Co. Redmond, WA)
Time Frame: 3 months after start of first intervention (Baseline to 3 months)
Population: The analyses included only subjects who completed all visits
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Number analyzed (Participants) | 39 | 41
unitless | -0.32 (0.96) | 0.09 (0.68)

2. Primary Outcome: Change in Vascular Function and Cardiometabolic Risk as Measured by Left CAVI at Month 8
Description: as for outcome 1
Time Frame: 3 months after start of second intervention (5 months to 8 months)
Population: The analyses included only subjects who completed all visits
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Number analyzed (Participants) | 38 | 36
unitless | -0.29 (0.55) | -0.07 (0.63)

3. Primary Outcome: Change in Vascular Function and Cardiometabolic Risk as Measured by Right CAVI at Month 3
Description: as for outcome 1
Time Frame: 3 months after start of first intervention (Baseline to 3 months)
Population: The analyses included only subjects who completed all visits
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Number analyzed (Participants) | 39 | 41
unitless | -0.42 (0.88) | 0.12 (0.65)

4. Primary Outcome: Change in Vascular Function and Cardiometabolic Risk as Measured by Right CAVI at Month 8
Description: as for outcome 1
Time Frame: 3 months after start of second intervention (5 months to 8 months)
Population: The analyses included only subjects who completed all visits
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Number analyzed (Participants) | 38 | 36
unitless | -0.26 (0.61) | -0.08 (0.71)

5. Primary Outcome: Change in Vascular Function and Cardiometabolic Risk as Measured by PWV at Month 3
Description: Change in vascular function using non-invasive vascular tests, measuring vascular compliance -Pulse, wave, velocity (PWV).
  The central aortic pressure PWV was determined by using the pressure tonometer and an EKG signal was used simultaneously to visualize ventricular-vascular interactions. It increases with atherosclerosis progression. Central aortic BP and stiffness were quantified using SphygmoCor CP system (AtCor Medical Pty Ltd.; New South Wales, Australia).
Time Frame: 3 months after start of first intervention (Baseline to 3 months)
Population: The analyses included only subjects who completed all visits
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Number analyzed (Participants) | 39 | 41
m/s | -0.31 (2.06) | 0.03 (2.03)

6. Primary Outcome: Change in Vascular Function and Cardiometabolic Risk as Measured by PWV at Month 8
Description: as for outcome 5
Time Frame: 3 months after start of second intervention (5 months to 8 months)
Population: The analyses included only subjects who completed all visits
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Number analyzed (Participants) | 38 | 36
m/s | -0.31 (1.86) | -0.25 (0.94)

7. Primary Outcome: Change in Vascular Function and Cardiometabolic Risk as Measured by RHI at Month 3
Description: Change in vascular function using non-invasive vascular tests, measuring vascular compliance -Reactive hyperemia index (RHI).
  RHI is a measure of endothelial dysfunction using noninvasive peripheral arterial tonometry (PAT). It is a ratio of the post-to-pre occlusion PAT amplitude of the tested arm, divided by the post-to-pre occlusion ratio of the control arm. RHI less than 1.67 is considered sign of endothelial dysfunction and RHI equal to or greater than 1.67 is considered normal function. The possible range of scores is 1 to 3. Increasing score indicates the improvement of coronary endothelial function
Time Frame: 3 months after start of first intervention (Baseline to 3 months)
Population: The analyses included only subjects who completed all visits
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Number analyzed (Participants) | 39 | 41
ratio | 0.07 (0.35) | 0.02 (0.48)

8. Primary Outcome: Change in Vascular Function and Cardiometabolic Risk as Measured by RHI at Month 8
Description: as for outcome 7
Time Frame: 3 months after start of second intervention (5 months to 8 months)
Population: The analyses included only subjects who completed all visits
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Number analyzed (Participants) | 38 | 36
ratio | -0.05 (0.35) | 0.02 (0.36)

9. Primary Outcome: Effect of Pioglitazone on Vascular Inflammation and Cardiometabolic Risk as Measured by TBR Value at Month 3
Description: Change in vascular inflammation using non-invasive vascular test, measuring changes in target to blood pool ratio (TBR) value by positron emission tomography (PET) computerized tomography (CT). The higher the value, the higher the degree of vascular inflammation.
Time Frame: 3 months after start of first intervention (Baseline to 3 months)
Population: The analyses included only subjects who completed all visits
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pioglitazone, Then Placebo | Placebo, Then Pioglitazone
Number analyzed (Participants) | 15 | 15
ratio | 0.0337 (0.1991) | 0.0351 (0.2954)

ADVERSE EVENTS:
Time Frame: 8 months
Groups:
- Pioglitazone: Treatment with pioglitazone up to 45 mg orally daily for three months.
- Placebo: Treatment with placebo orally daily for 3 months.
Arm/Group | Pioglitazone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 1/77 | 5/77
Other Adverse Events (participants affected / at risk) | 33/77 | 33/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=77) | Placebo (N=77)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 | 1 (1)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=77) | Placebo (N=77)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0
Osler's nodes (Cardiac disorders) | 0 | 1 (1)
Tachycardia (Cardiac disorders) | 0 | 1 (1)
Dry eye (Eye disorders) | 0 | 1 (1)
Episcleritis (Eye disorders) | 1 (1) | 0
Lacrimation increased (Eye disorders) | 1 (1) | 0
Vision blurred (Eye disorders) | 0 | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0
Gastritis (Gastrointestinal disorders) | 2 (2) | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Oral pain (Gastrointestinal disorders) | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0
Administration site pain (General disorders) | 0 | 1 (1)
Fatigue (General disorders) | 5 (5) | 1 (1)
Feeling cold (General disorders) | 0 | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0
Localised oedema (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 | 1 (1)
Peripheral swelling (General disorders) | 0 | 1 (1)
Gastritis viral (Infections and infestations) | 1 (1) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0
Influenza (Infections and infestations) | 0 | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 10 (11)
Urinary tract infection (Infections and infestations) | 1 (1) | 9 (10)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0
Exposure to allergen (Injury, poisoning and procedural complications) | 0 | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0
Alanine aminotransferase increased (Investigations) | 5 (5) | 0
Aspartate aminotransferase increased (Investigations) | 2 (3) | 3 (3)
Biopsy lymph gland (Investigations) | 1 (1) | 0
Blood bicarbonate decreased (Investigations) | 1 (2) | 0
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood urea increased (Investigations) | 0 | 1 (1)
Cardiac murmur (Investigations) | 3 (3) | 0
Computerised tomogram abnormal (Investigations) | 1 (1) | 0
Computerised tomogram coronary artery abnormal (Investigations) | 1 (1) | 0
Helicobacter test positive (Investigations) | 1 (1) | 0
International normalised ratio increased (Investigations) | 0 | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2) | 1 (2)
Platelet count decreased (Investigations) | 2 (2) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 0
Weight increased (Investigations) | 3 (3) | 0
White blood cell count decreased (Investigations) | 7 (8) | 1 (1)
Anorexia nervosa (Metabolism and nutrition disorders) | 1 (1) | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Chills (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0
Dizziness (Nervous system disorders) | 4 (5) | 7 (7)
Headache (Nervous system disorders) | 2 (2) | 7 (8)
Memory impairment (Nervous system disorders) | 1 (1) | 0
Numbness (Nervous system disorders) | 1 (1) | 0
Paraesthesia (Nervous system disorders) | 2 (3) | 0
Presyncope (Nervous system disorders) | 0 | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 0 | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0
Cystitis (Renal and urinary disorders) | 0 | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 0
Fluid retention (Renal and urinary disorders) | 1 (1) | 0
Micturition disorder (Renal and urinary disorders) | 2 (2) | 0
Nocturia (Renal and urinary disorders) | 0 | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 | 1 (1)
Galactorrhoea (Reproductive system and breast disorders) | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT02338999/Prot_SAP_000.pdf